CLINICAL TRIAL: NCT00487708
Title: An Open-Label, Phase II Dose Titration Study of ACZ885 (Human Anti-IL-1β Monoclonal Antibody) to Assess the Clinical Efficacy, Safety, Pharmacokinetics and Pharmacodynamics in Patients With NALP3 Mutations
Brief Title: Safety, Efficacy, Pharmacokinetics, Pharmacodynamics of ACZ885 in Patients With NALP3 Mutations and Clinical Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885A2102
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: NALP3 Mutation
Keywords: ACZ885; NALP3 mutations; Interleukin-1beta; Muckle-Wells Syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): ACZ885
  Interventions: Drug: canakinumab

INTERVENTIONS:
Drug: canakinumab

SUMMARY:
This study will investigate the clinical efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of ACZ885, administered intravenously and subcutaneously to patients with NALP3 mutations whose clinical symptoms are either untreated or insufficiently treated and require medical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4 to 75 years (inclusive)
* Body weight ≥ 12 kg and < 100 kg.
* Females of child-bearing potential must have a negative pregnancy test. Additional birth control details to be provided at screening.
* Documented molecular diagnosis of NALP3 mutations and clinical symptoms that are either untreated or insufficiently treated and require medical intervention.
* Patients under anakinra therapy or any other IL-1 blocking therapy, whose clinical symptoms improved under treatment and are willing to discontinue that therapy until a relapse becomes evident.
* Patients with a very severe characteristics requiring oral prednisone are eligible if the dose is stable (≤ 0.4 mg/kg/day or ≤ 20 mg/day, whichever is lower) for at least 1 week prior to the screening visit. Steroid therapy may be tapered during treatment with ACZ885 at the discretion of the investigator.
* Parents' or legal guardian's written informed consent (patient's informed consent for ≥ 18 years of age) and child's assent, if appropriate, are required prior to study participation.

Exclusion Criteria:

* Participation in any clinical trial investigation (except trials with anakinra) within 4 weeks prior to dosing or longer per local regulation
* Antiinflammatory therapy with colchicine, chlorambucil, dapsone, azathioprine, mycophenolate mofetil, within 3 weeks prior to dosing. Therapeutic antibodies (e.g. anti-TNF-alpha antibodies) must be discontinued at least 60 days before dosing.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* A past personal or close family medical history of clinically significant ECG abnormalities or prolonged QT-interval syndrome.
* History of

  * Immunocompromise, including a positive HIV result.
  * Positive Hepatitis B surface antigen or Hepatitis C test result.
  * Drug or alcohol abuse within the 12 months prior to dosing.
  * Tuberculosis.
  * Renal transplant.
  * Evidence of lymphoma.
* Active medical condition preventing participation in the study such as infection, poorly controlled diabetes etc.
* No live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Response to treatment and time to relapse after ACZ885 administration according to monthly investigator's clinical assessments, laboratory monitoring, and patient diaries. | Every month

SECONDARY OUTCOMES:
Assessment of safety,tolerability and immunogenicity of ACZ885 at each clinical visit. Evaluation of ACZ885 PK and PD at each clinical visit Evaluate efficacy towards hearing loss(every 4 months),kidney function (every 4 months),neurological symptoms | Every month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (10):
- Novartis Investigator Site, Lille, France
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Dresden
  - Novartis Investigator Site, Heidelberg
  - Novartis Investigator Site, Marburg
  - Novartis investigative site, Nuremberg
  - Novartis Investigator Site, Tübingen
- Novartis Investigator Site, New Dehli, India
- Novartis Investigator Site, Oviedo, Spain
- Novartis Investigative site, London, United Kingdom

REFERENCES:
- [Derived] Kuemmerle-Deschner JB, Ramos E, Blank N, Roesler J, Felix SD, Jung T, Stricker K, Chakraborty A, Tannenbaum S, Wright AM, Rordorf C. Canakinumab (ACZ885, a fully human IgG1 anti-IL-1beta mAb) induces sustained remission in pediatric patients with cryopyrin-associated periodic syndrome (CAPS). Arthritis Res Ther. 2011 Feb 28;13(1):R34. doi: 10.1186/ar3266. PMID 21356079